CLINICAL TRIAL: NCT01406093
Title: Early- and Late-onset Candidemia: A Retrospective Study
Brief Title: Early- and Late-onset Candidemia
Status: Completed | Type: Observational
Sponsor: Giovanni Di Perri (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Giovanni Di Perri, Early- and Late-onset Candidemia, University of Turin, Italy
Organization: University of Turin, Italy (Other)
Other Study IDs: EOC1-11
Record Dates: First submitted 2011-07-28; First posted 2011-07-29 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Candidemia
Keywords: Candidemia; Early-onset; Late-onset; Health-care associated; Nosocomial
MeSH Terms: conditions — Candidemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Candidemia patients: Patients with diagnosis of candidemia

SUMMARY:
A timing diagnosis of candidemia is as important as the correct choice of empiric or targeted antifungal therapy. In the last years a growing body of knowledge has better characterized health-care associated (HCA) infections, which have been described in 2002 in outpatients with MRSA bloodstream infections. So far there is no compelling evidence that patients with HCA infections may develop candidemia before the usual timing of around 20-25 days after admission. Risk factors associated with HCA infections are represented by admission from long term chronic care facilities (LTCF), haemodialysis, previous admission or parenteral broad spectrum antibiotics. There are few data HCA features and early onset candidemias in the published literature.

In this proposal, the investigators aim at studying early-onset candidemia in a retrospective study in one of the largest referral hospital in Italy with a consistent range of specialties ranging (bone marrow transplant, solid organ transplant, immunosuppressed patients, ICU, complex surgery). The investigators speculate that patients with candidemia diagnosed within 10 days (early-onset) by the admission have different risk factors and prognosis of those with a late diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Candidemia diagnosed with positive blood culture either from a peripheral vein or CVC

Exclusion Criteria:

* Candida isolated from a removed CVC tip will not be considered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The selection of patients for inclusion will be based on microbiological data (with suscesptibilty patterns of the various antifungals) extracted from the computerized archive with search for Candida spp. and "blood" either peripheral or from a central venous catheter. Candida isolated from a removed CVC tip will not be considered. The candidemia will also be defined early or late based on the time elapsed between hospital admission and diagnosis (≤ 10 days early, > 10 days late candidemia).
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2011-05; Primary Completion 2012-02 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Mortality | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Di Perri, MD, PhD, Principal Investigator — University of Turin, Italy; Francesco G De Rosa, MD, Study Chair — University of Turin, Italy
Locations (1):
- Hospital San Giovanni Battista - Molinette, Torino, Italy